CLINICAL TRIAL: NCT00415519
Title: An Exploratory Study of MCI-186 for Treatment of Amyotrophic Lateral Sclerosis (Severity Classification III) in Double-Blind, Parallel-Group, Placebo-Controlled Manner
Brief Title: Efficacy and Safety Study of MCI-186 for Treatment of Amyotrophic Lateral Sclerosis (ALS) Who Met Severity Classification III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI186-18
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic lateral sclerosis; free radical scavenger
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MCI-186
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo of MCI-186

INTERVENTIONS:
Drug: MCI-186 — Two ampoules (60 mg) of MCI-186 injection are intravenously administered once a day, for successive 14 days, followed by 14 days observation period (first cycle). Then treatment (10 days' administration during 14 days) - observation (14 days) cycle is repeated five times (2nd-6th cycles).
  Other Names: Edaravone; Radicut
  Arms: 1
Drug: Placebo of MCI-186 — Two ampoules of Placebo injection are intravenously administered once a day, for successive 14 days, followed by 14 days observation period (first cycle). Then treatment (10 days' administration during 14 days) - observation (14 days) cycle is repeated five times (2nd-6th cycles).
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate the efficacy of 60mg of MCI-186 via intravenous drip once a day in patients with ALS whose severity is classified as grade III, based on the changes in the revised ALS functional rating scale (ALSFRS-R) scores after 24 weeks administration in double-blind, placebo-controlled manner. And in addition, this study will be performed to examine the safety of MCI-186 to ALS patients who met severity classification III.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are defined as "definite ALS," "probable ALS" or "probable-laboratory-supported ALS," met diagnostic criteria revised EL Escorial for Airlie House.
* Patients who cannot take at least one action of eating a meal, excreting, or moving with oneself alone, and need assistance in everyday life.
* Patients whose progress of the condition during 12 weeks before administration meet other requirements.

Exclusion Criteria:

* Patients judged to be inadequate to participate in this study by their physician, because those patients' general condition deteriorated to the point that they need to be hospitalized for severe hepatic disease, sever heart disease, sever renal disease and so on, or they need to be administered antibiotics to infection.
* Patients who complain the difficulty in breathing caused by deteriorating the respiratory function.
* Patients with such complications as Parkinson's disease, schizophrenia, dementia, renal failure, or other severe complication, and patients who have the anamnesis of hypersensitivity to edaravone.
* Pregnant, lactating, and probably pregnant patients, and patients who want to become pregnant, and patients who can not agree to contraception.
* Patients who have been administered other investigational products within 12 weeks before consent, or who are participating in other clinical trials at present.
* In addition to the above exclusion criteria, patients judged to be inadequate to participate in this study by their physician.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koji Abe, professor, Principal Investigator — Graduate School of Medicine and Dentistry, Okayama University

REFERENCES:
- [Result] WRITING GROUP ON BEHALF OF THE EDARAVONE (MCI-186) ALS 18 STUDY GROUP. Exploratory double-blind, parallel-group, placebo-controlled study of edaravone (MCI-186) in amyotrophic lateral sclerosis (Japan ALS severity classification: Grade 3, requiring assistance for eating, excretion or ambulation). Amyotroph Lateral Scler Frontotemporal Degener. 2017 Oct;18(sup1):40-48. doi: 10.1080/21678421.2017.1361441. PMID 28872915

RESULTS

PARTICIPANT FLOW:
Groups:
- MCI-186: MCI-186 Injection 30 mg, 2 ampoules per treatment, once daily, intravenously infused over 60 min
- Placebo of MCI-186: MCI-186 Injection Placebo, 2 ampoules per treatment, once daily, intravenously infused over 60 min
Period: Overall Study
Arm/Group | MCI-186 | Placebo of MCI-186
Started | 13 | 12
Completed | 9 | 12
Not Completed | 4 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Patient's convenience | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCI-186 | Placebo of MCI-186 | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Revised ALS Functional Rating Scale (ALSFRS-R) Score in Full Analysis Set (FAS) Population at 24 Weeks
Description: No primary endpoint was used, because various exploratory analyses were performed.
  0=worst; 48=best
Time Frame: baseline and 24 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 13 | 12
units on a scale | -6.52 (1.78) | -6 (1.83)

2. Primary Outcome: Death or a Specified State of Disease Progression
Description: No primary endpoint was used, because various exploratory analyses were performed.
  Any of "death, disability of independent ambulation, loss of upper arm function, tracheotomy, use of respirator, and use of tube feeding" was defined as an event.
Time Frame: 24 weeks
Measure: Number; unit: events
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 13 | 12
events
  death | 1 | 0
  disability of independent ambulation | 4 | 2
  loss of upper arm function | 1 | 2
  tracheotomy | 0 | 0
  use of respirator | 0 | 0
  use of tube feeding | 1 | 0

3. Primary Outcome: Change From Baseline in % Forced Vital Capacity (%FVC) in Full Analysis Set (FAS) Population at 24 Weeks
Description: No primary endpoint was used, because various exploratory analyses were performed.
Time Frame: baseline and 24 weeks
Population: "1 patient with missing value at baseline" was excluded from the FAS in the MCI-186 group.
Measure: Least Squares Mean (Standard Error); unit: percentage of FVC
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 12 | 12
percentage of FVC | -18.75 (4.58) | -15.69 (4.58)

4. Primary Outcome: Percentage of Participants With Adverse Events
Description: No primary endpoint was used, because various exploratory analyses were performed.
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 13 | 12
percentage of participants | 92.3 | 100

5. Primary Outcome: Percentage of Participants With Adverse Drug Reactions
Description: No primary endpoint was used, because various exploratory analyses were performed.
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 13 | 12
percentage of participants | 23.1 | 8.3

6. Primary Outcome: The Percentage of Participants With an Abnormal Change in Laboratory Tests That Occurred in More Than Two Patients
Description: No primary endpoint was used, because various exploratory analyses were performed.
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 13 | 12
percentage of participants
  White blood cell count (WBC) | 23.1 | 8.3
  Other laboratory tests except for WBC | 0 | 0

7. Primary Outcome: Percentage of Participants With Abnormal Changes in Sensory Examinations
Description: No primary endpoint was used, because various exploratory analyses were performed.
Time Frame: 24 weeks
Population: A note:
  Each three patients of both groups did not have data to Staggering due to data missing. Therefore, concerning staggering, the number of participants analysed are 10 in the MCI-186 group and 9 in the placebo of MCI-186 group.
Measure: Number; unit: percentage of participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 13 | 12
percentage of participants
  Numbness | 0 | 0
  Staggering: number analyzed (Participants) | 10 | 9
  Staggering | 10 | 0
  Vibratory sensation | 0 | 0

ADVERSE EVENTS:
Arm/Group | MCI-186 | Placebo of MCI-186
Serious Adverse Events (participants affected / at risk) | 3/13 | 2/12
Other Adverse Events (participants affected / at risk) | 12/13 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-186 (N=13) | Placebo of MCI-186 (N=12)
Dysphagia (Gastrointestinal disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-186 (N=13) | Placebo of MCI-186 (N=12)
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dyschezia (Gastrointestinal disorders) | 0 | 3
Gingivitis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 3
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Abasia (General disorders) | 0 | 1
Feeling cold (General disorders) | 1 | 0
Gait disturbance (General disorders) | 3 | 1
Impaired healing (General disorders) | 1 | 0
Thirst (General disorders) | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2
Oral herpes (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 2
Blood urine present (Investigations) | 0 | 1
Glucose urine present (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 2
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other